CLINICAL TRIAL: NCT01704950
Title: Clinical Outcome of Defect Reconstruction Using IDRT Single Layer : Results From a Prospective Multicentric Trial
Status: Completed | Type: Observational
Sponsor: Integra LifeSciences Services (Industry)
Responsible Party: Sponsor
Other Study IDs: RECON-EMEA-11
Record Dates: First submitted 2012-10-09; First posted 2012-10-12 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Traumatic Wound; Reconstruction Wound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to provide data and the guidelines for the use of IDRT SL in small wounds, acute and chronic (less than 6 months), showing the benefits and the easy to use of this product as a one stage procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient with 1 traumatic wound (burns included) or 1 reconstruction wound (oncological wounds included)
* Patients for whom the surgeon has recommended that an INTEGRA® SL matrix be implanted (even if the patient is not taking part in the study) with a Split Thickness Skin Graft in the same operating procedure
* Wound treated with only one layer of a maximum size 10cm*12.5cm

Exclusion Criteria:

* Immunosuppressed patient
* Chronic wound (with no healing since 6 months)
* Addition of any substances (growth factor, stem cells,…) in the IDRT SL during the surgery
* Patient with a corticoid treatment with a daily dose greater than 5 mg
* Patients whose life expectancy is less than 12 months
* Patients whose mental health or health condition (Visual deficiency, Alzheimers…) would compromise completion of the self-evaluation questionnaires
* Patient with an hypersensitivity to bovine collagen, chondroitin
* Patient with clinical signs of infection (fever, pain, colour, swelling,…) and for whom the investigator diagnosed infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Global population
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2013-02; Primary Completion 2014-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Rate of graft take | Day 15 after the surgery
  the mean percentage of healing expected at Day 15 after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Stefanos Papadopoulos, Principal Investigator — General State Hospital of Athens, "G. Gennimatas"
Locations (4):
- St Josef Hospital, Bochum, Germany
- General State Hospital of Athens, "G. Gennimatas" - Department of Plastic Surgery-Microsurgery and Burn Center, Athens, Greece
- University Hospital "S. Maria della Misericordia" - Plastic Surgery and Burn Center, Udine, Italy
- Queen Elizabeth Hospital - Burn and Plastic Surgery, Birmingham, United Kingdom